CLINICAL TRIAL: NCT05695131
Title: Clinical Implementation, Feasibility, & Validation of the Virtual Reality Delivered GlenxRose Speech-Language Therapies to Improve Patient Adherence and Treatment Outcomes
Brief Title: Clinical Feasibility & Validation of the Virtual Reality GlenxRose Speech-Language Therapies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00126403
Record Dates: First submitted 2023-01-04; First posted 2023-01-23 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Vocal Cord Dysfunction; Speech Disorders
Keywords: Vocal; Speech; Speech-Language Pathology; Virtual Reality; VR
MeSH Terms: conditions — Vocal Cord Dysfunction; Speech Disorders; Speech

STUDY DESIGN:
Intervention Model Description: Study 1: Single-Subject Experimental Design Studies will be Implemented (A-B Design) Study 2: Feasibility randomized controlled trial (control and intervention groups)
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be masked to group allocation (VR-delivered therapy + standard care, or traditional standard care alone). Participants will be asked by a research assistant not to reveal details of the group allocation prior to assessments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Delivered Therapy + Standard Clinical Care (Experimental): The GlenXRose virtual reality therapies will be delivered to participants using a head-mounted device to allow vocal therapy and practice. Participants will also receive routine clinical care provided by speech-language pathologists.
  Interventions: Device: GlenXRose Virtual Reality Speech Therapies
- Standard Clinical Care (No Intervention): Participants will receive routine clinical care provided by speech-language pathologists.

INTERVENTIONS:
Device: GlenXRose Virtual Reality Speech Therapies — Speech therapies for vocal cord disorders have been developed for virtual reality implementation. These include various games to interact with in a virtual environment while conducting rehabilitation therapy, in addition to educational visualizations
  Arms: Virtual Reality Delivered Therapy + Standard Clinical Care

SUMMARY:
Factors related to successful rehabilitation are often directly related to adherence; for instance, dosage, frequency, and intensity can burden the patient regarding time and motivational factors. Furthermore, surrounding salience, patients may lose interest or find an intervention boring after a few sessions. It is well documented that nonadherence not only impacts rehabilitation for the patient but can also further prolong treatment, and increase hospital and clinician costs, in addition to a higher prevalence of future comorbidities. Therefore, strategies that improve patient adherence can significantly help optimize patient care and treatment outcomes.

One avenue to increase patient adherence is through the gamification of rehabilitation therapies using virtual reality (VR). Gamification of rehabilitation therapy can make mass practice required in rehabilitation therapies seemingly fun and more personally engaging for the patient. Additionally, the immersive experience achieved through VR can further promote salience and be customizable to individual patient requirements. As VR systems are now highly portable and relatively simple to utilize, they can provide an excellent opportunity to continue rehabilitation practice on the home front. Overall, the VR gamification of rehabilitation may increase adherence by shifting patients' perspectives of therapy as tedious, boring, or a hassle, to a fun and engaging game that ultimately helps their recovery processes.

The GlenXRose VR-delivered speech-language therapies (Cognitive Projections Lab, University of Alberta) have been developed and piloted in collaboration with the Glenrose Rehabilitation Hospital with the overall goal of increasing patient adherence, treatment outcomes, and satisfaction with vocal therapy. The proposed studies are to investigate the feasibility of implementing this technology in routine clinical care (specific to voice disorders), obtaining clinician feedback, examining associated financial costs, and continuing to examine the effect of the GlenXRose VR speech-language therapies on patient adherence and clinical outcomes, compared to traditional clinical care.

DETAILED DESCRIPTION:
Nonadherence to Speech-Language rehabilitation can result in suboptimal vocal recovery or compensation methods while impacting the quality of life and further burdening the healthcare system. In addition to traditional face-to-face voice therapy, many patients are further given daily voice exercises to practice at home. It is estimated that 38-74% of patients are nonadherent to voice therapies (Ebersole et al., 2018); with such a large prevalence, opportunities to prevent and mitigate nonadherence to voice therapy can significantly promote clinical/functional outcomes. In a recent meta-analysis, it is reported that methods increasing adherence to speech-language rehabilitation further promote home practice (Bartlett et al., 2022). One identified method of promise includes technological approaches (Bartlett et al., 2022) such as the GlenXRose VR Speech-Language therapies (VR-SLP).

Purpose & Objective: The GlenXRose VR-SLP program, developed by the Cognitive Projections lab at the University of Alberta in collaboration with the Glenrose Rehabilitation Hospital, provides patients with gamified vocal exercises, therapies, and education delivered through immersive virtual reality. With the degree of VR portability, patients will be able to take the equipment home to facilitate at-home vocal practice.

The objective of these studies is to examine the feasibility of implementing the previously developed GlenXRose VR Speech Language therapies (VR-SLP) to routine clinical care delivered by Speech-Language Pathologists to patients with vocal cord disorders. The variables of patient adherence to treatment as well as preliminary effects on vocal measurements (Voice Handicapped Index - 10; Acoustic Analysis of Voice) will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Adults receiving speech-language therapy at the Glenrose Rehabilitation Hospital (Edmonton, AB, Canada; Alberta Health Services)
* Presence of a speech disorder
* Proficiency in English
* Able to provide signed informed consent to participate in the study

Exclusion Criteria:

* Severe cognitive impairments and/or behavioural impairments
* Communication disorders that impact comprehension of verbal commands and understanding of scale used in the study
* Previous history of neurological or psychiatric disorder
* Substance use disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Frequency and Treatment Adherence Rates | Up to 12 Weeks
  Reported Frequency of Rehabilitation Therapy
Change in Generalization | Up to 12 Weeks
  Self-reported time using voice production techniques
Change in Compliance Rate | Up to 12 Weeks
  Self-reported time (using a visual analog scale)
Change in Voice Handicap Index - 10 | Up to 12 Weeks
  Quantification of participant reported perspectives of voice impairment(s)
Change in Acoustic Analysis of Voice | Up to 12 Weeks
  Conducted by Registered Speech-Language Pathologists (as part of standard care)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Rios Rincon, PhD, R.OT, Principal Investigator — University of Alberta; Antonio Miguel Cruz, DrSc, Study Chair — University of Alberta; James Raso, MASc, Study Chair — Glenrose Rehabilitation Hospital, Alberta Health Services
Locations (1):
- Glenrose Rehabilitation Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosen CA, Lee AS, Osborne J, Zullo T, Murry T. Development and validation of the voice handicap index-10. Laryngoscope. 2004 Sep;114(9):1549-56. doi: 10.1097/00005537-200409000-00009. PMID 15475780
- [Background] Bartlett RS, Carpenter AM, Chapman LK. A Systematic Review of Adherence Strategies for Adult Populations in Speech-Language Pathology Treatment. Am J Speech Lang Pathol. 2022 May 10;31(3):1501-1516. doi: 10.1044/2022_AJSLP-21-00255. Epub 2022 Mar 23. PMID 35320678
- [Background] Ebersole B, Soni RS, Moran K, Lango M, Devarajan K, Jamal N. The Role of Occupational Voice Demand and Patient-Rated Impairment in Predicting Voice Therapy Adherence. J Voice. 2018 May;32(3):325-331. doi: 10.1016/j.jvoice.2017.06.002. Epub 2017 Jul 11. PMID 28709763
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. Pilot Feasibility Stud. 2016 Oct 21;2:64. doi: 10.1186/s40814-016-0105-8. eCollection 2016. PMID 27965879